CLINICAL TRIAL: NCT03134703
Title: Methadone Demonstration Project With Neonatal Intensive Care Unit Infants Diagnosed With Neonatal Abstinence Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Johns Hopkins All Children's Hospital (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00107690
Record Dates: First submitted 2017-03-03; First posted 2017-05-01 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Methadone; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone Treatment Group (Experimental): NAS infants treated for withdrawal symptoms with methadone
  Interventions: Drug: Methadone
- Comparison Group (Active Comparator): NAS infants treated for withdrawal symptoms with morphine (standard of care at Johns Hopkins All Children's Hospital)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Infants in the Methadone Treatment Group will receive the study drug, methadone, instead of morphine to treat withdrawal symptoms from Neonatal Abstinence Syndrome (NAS)
  Arms: Methadone Treatment Group
Drug: Morphine — Infants in the Comparison Group will receive standard of care narcotic (morphine) to treat withdrawal symptoms from Neonatal Abstinence Syndrome (NAS)
  Arms: Comparison Group

SUMMARY:
This is a non-randomized, un-blinded feasibility study project comparing the Length of Stay (LOS) of Neonatal Intensive Care Unit (NICU) infants diagnosed with Neonatal Abstinence Syndrome (NAS) treated with methadone with historical data and a comparison group of NICU NAS infants treated with a different narcotic agent.

DETAILED DESCRIPTION:
For the time frame July 1, 2013 through September 30, 2014, 300 infants with NAS have been cared for in the JHACH NICU with an average length of stay of 30 days. Such a prolonged length of stay has a negative impact on maternal/infant bonding. In addition, infants suffering from NAS have poor regulatory mechanisms and are invariably hard to care for and difficult to console, and they provide an emotional challenge to their caretakers. This challenge becomes even more significant when the caretaker is the mother who is suffering from addiction and is already emotionally compromised by feelings of depression, anxiety, guilt or insecurity. Attachment is an ongoing process and the quality of the relationship between mother and her infant directly influences the structure of the child's affective ties and overall organization of responses to environment. This mother-infant bond sets the stage for understanding and identifying the infant's needs and reciprocal parental response to those needs. Maternal emotional unavailability has potentially serious effects on the long term mother-child relationship, and on the child's development.

This project provides a novel approach and an alternative care plan for infants with NAS. It is funded by the State of Florida and allows to: 1) educate and empower a specified population of mothers who are undergoing institutionalized rehabilitation and whose infant needs treatment for NAS; 2) safely transition the infants home for final wean of their pharmacologic treatment; 3) provide regular developmental follow up for these infants through our NICU follow up clinic, hence identifying and quickly responding to neuro-developmental delays.

ELIGIBILITY:
Methadone Treatment Group:

Inclusion criteria:

1. Baby is diagnosed with neonatal abstinence syndrome;
2. Mother under the care of Operation PAR;
3. Mother resides in Pinellas or Pasco county at the time of enrollment and is expected to throughout the infant's methadone treatment period;
4. Mother has been deemed by PAR officials as being compliant with the detoxification program;
5. Mother has completed induction methadone treatment and has had no changes in medication dosage of 10% or greater in the two weeks preceding delivery;
6. Mother has been prescreened and deemed adequate candidate by the demonstration project team members;
7. No known concerns from Florida Department of Children and Families regarding the infant's ability to return to the home;
8. Newborns ≥ 37 0/7 weeks gestation;
9. Newborns transferred to JHACH within 72 hours from birth;
10. Newborns ≥ 2.5 kg weight at birth;
11. Informed parental consent.

Exclusion Criteria:

1. Major congenital anomalies;
2. Major concomitant medical illness including planned antibiotic treatment for greater than 3 days or NPO status;
3. Infants who are being placed for adoption;
4. Infants in significant pain requiring narcotic medication for comfort (for example those with a fracture);
5. Infants whose maternal UDS at the time of delivery is positive for any other drug of abuse beside opiates.
6. Mother with hearing or language impairment

Comparison Group:

Inclusion Criteria:

1. Baby is diagnosed with neonatal abstinence syndrome;
2. Newborns ≥ 37 0/7 weeks gestation;
3. Newborns transferred to JHACH within 72 hours from birth;
4. Newborns ≥ 2.5 kg weight at birth;
5. Informed parental consent.

Exclusion Criteria:

1. Infant not requiring pharmacologic treatment for NAS;
2. Major congenital anomalies;
3. Major concomitant medical illness including planned antibiotic treatment for greater than 3 days or NPO status;
4. Infants who are being placed for adoption;
5. Infants in significant pain requiring narcotic medication for comfort (for example those with a fracture);
6. Mother with hearing or language impairment;
7. Infants known upon admission who will be placed into state custody or sheltered.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Brooks, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone Treatment Group | Comparison Group
Started | 6 | 5
Completed | 0 | 3
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone Treatment Group | Comparison Group | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: Days] | 1.5 [1 to 2] | 10.4 [5 to 20] | 5.5 [1 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay (LOS)
Description: Compare the LOS of Neonatal Intensive Care Unit (NICU) infants with Neonatal Abstinence Syndrome (NAS) treated with methadone with historical data and a comparison group of NICU NAS infants treated with a different narcotic agent.
Time Frame: 25 days
Population: Study closed prematurely due to poor accrual. There were 3 screen fails (did not receive study drug) in the methadone treatment group, therefore LOS was not calculated for those participants.
Measure: Mean (Full Range); unit: days
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 3 | 5
days | 11.3 [9 to 15] | 16.2 [6 to 25]

2. Secondary Outcome: Maternal Bonding Measured With The Postpartum Bonding Questionnaire (PBQ)
Description: The Postpartum Bonding Questionnaire (PBQ) is a self-rating questionnaire designed to detect disorders of the mother-infant relationship. The questionnaire has 25 statements, each with six alternative responses ranging from 0 (always) to 5 (never). For the PBQ, scores are summated for each factor, with a high score indicating concern for bonding. The PBQ yields a total score between 0 to 125. Positive responses are scored from 0 ('always') to 5 ('never'). Negative responses, are scored from 5 ('always') to 0 ('never').
  Factor 1 (impaired bonding) is based on 12 questions, with a score range 0-60 (0-11=normal; 12 & above=high).
  Factor 2 (rejection & anger) is based on 7 questions with a score range 0-35 (0-16=normal; 17 & above=high).
  Factor 3 (anxiety about care) is based on 4 questions with a score range 0-20 (0-9=normal; 10 & above =high).
  Factor 4 (risk of abuse) is based on 2 questions, with a score range 0-10 (0-2=normal; 3 & above =high).
Time Frame: inpatient and at 6-8 weeks of age
Population: Data analysis was not completed. Results shown below are means for each group, note that many participants replied on the extremes of the answer range (e.g. always or never), which yields very low total scores for each factor.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 5 | 5
score on a scale
  Factor 1 inpatient | 0 [0 to 0] | 0.4 [0 to 2]
  Factor 2 inpatient | 0 [0 to 0] | 0 [0 to 0]
  Factor 3 inpatient | 0.6 [0 to 1] | 1 [0 to 2]
  Factor 4 inpatient | 0 [0 to 0] | 0 [0 to 0]
  Factor 1 6-8 weeks: number analyzed (Participants) | 1 | 2
  Factor 1 6-8 weeks | 1 [1 to 1] | 0.5 [0 to 1]
  Factor 2 6-8 weeks: number analyzed (Participants) | 1 | 2
  Factor 2 6-8 weeks | 0 [0 to 0] | 1 [0 to 2]
  Factor 3 6-8 weeks: number analyzed (Participants) | 1 | 2
  Factor 3 6-8 weeks | 0 [0 to 0] | 2.5 [2 to 3]
  Factor 4 6-8 weeks: number analyzed (Participants) | 1 | 2
  Factor 4 6-8 weeks | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Maternal Depression Measured With The Edinburgh Postnatal Depression Scale (EPDS)
Description: The Edinburgh Postnatal Depression Scale (EPDS) was developed for screening postpartum women in outpatient, home visiting settings, or at the 6-8 week postpartum examination. The EPDS is a 10-item questionnaire with responses scored 0, 1, 2, or 3 according to increased severity of the symptom. The maximum total score is 30 while the minimum score is 0. A score of 10 or greater, as well as any answer choice other than "never" on question #10 (suicidal thoughts) of the EPDS are indicative of depressive symptomatology.
Time Frame: While inpatient and at 6-8 weeks of age
Population: Data analysis was not completed. Results shown below are average scores on the EPDS scale for each group. 9 participants completed the EPDS while in patient, and 4 participants completed the questionnaire at the 6-8 weeks time point.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 4 | 5
score on a scale
  EPDS inpatient | 0.3 [0 to 1] | 7.2 [1 to 20]
  EPDS 6-8 weeks: number analyzed (Participants) | 1 | 3
  EPDS 6-8 weeks | 10 [10 to 10] | 5.3 [1 to 14]

4. Secondary Outcome: Readmission to Hospital
Description: Number of hospital readmissions
Time Frame: Within 30 days of discharge
Population: Readmissions to the hospital within 30 days for NAS-related reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

5. Secondary Outcome: Breast Milk
Description: Compare the incidence of providing breast milk (> 50% of nutritional needs) at 30 days of age between methadone treated and non-treated infants
Time Frame: 30 days of age
Population: Study closed prematurely due to poor accrual and no analysis was completed. Incidence of providing breast milk at 30 days was not collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Infant Development
Description: Assess the age appropriate infant development at 4, 8 and 12 months of age among the methadone treatment group using the Ages and Stages-based questionnaires (ASQ). The questionnaires are screening tools designed to identify infants at risk for developmental delays through caregivers' provision of quantitative information regarding their infant's development. In the ASQ, higher scores indicate more positive outcomes. The ASQ covers 5 areas of development: communication, gross motor, fine motor, problem solving, and personal-social. Scores for each area should fall between 0-60.
  Scoring:
  0-30 = further assessment with a professional may be needed 30-40 = learning activities & monitoring are indicated 45-60 = child development appears to be on schedule
Time Frame: 4, 8 and 12 months of age
Population: Infant development assessed only on those participants who received study drug (methadone arm). 3 participants completed the ASQ at 4 months, 1 participant at 8 months, and 1 participant at 12 months.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 3 | 0
score on a scale
  Communication at 4m | 51.7 [45 to 60] |
  Gross motor at 4m | 56.7 [50 to 60] |
  Fine motor at 4m | 56.7 [55 to 60] |
  Problem solving at 4m | 56.7 [50 to 60] |
  Personal-social at 4m | 60 [60 to 60] |
  Communication at 8m: number analyzed (Participants) | 1 | 0
  Communication at 8m | 60 [60 to 60] |
  Gross motor at 8m: number analyzed (Participants) | 1 | 0
  Gross motor at 8m | 50 [50 to 50] |
  Fine motor at 8m: number analyzed (Participants) | 1 | 0
  Fine motor at 8m | 50 [50 to 50] |
  Problem solving at 8m: number analyzed (Participants) | 1 | 0
  Problem solving at 8m | 55 [55 to 55] |
  Personal-social at 8m: number analyzed (Participants) | 1 | 0
  Personal-social at 8m | 50 [50 to 50] |
  Communication at 12m: number analyzed (Participants) | 1 | 0
  Communication at 12m | 50 [50 to 50] |
  Gross motor at 12m: number analyzed (Participants) | 1 | 0
  Gross motor at 12m | 40 [40 to 40] |
  Fine motor at 12m: number analyzed (Participants) | 1 | 0
  Fine motor at 12m | 60 [60 to 60] |
  Problem solving at 12m: number analyzed (Participants) | 1 | 0
  Problem solving at 12m | 50 [50 to 50] |
  Personal-social at 12m: number analyzed (Participants) | 1 | 0
  Personal-social at 12m | 40 [40 to 40] |

7. Secondary Outcome: Screened vs. Eligible
Description: Determine the response percentage of mothers who are screened as eligible by PAR officials and who agree to participate in the demonstration project
Time Frame: After accrual of the first 50% of participants & after accrual of the second 50% of participants, and at completion of the trial.
Population: Study closed prematurely due to poor accrual and no analysis was completed. Response percentage was not collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Attrition Rate
Description: Assess the drop out percentage of mothers who agree to participate but do not follow through with home discharge for continued care
Time Frame: After accrual of the first 50% of participants, after accrual of the second 50% of participants, and at completion of the trial.
Population: Study closed prematurely due to poor accrual and no analysis was completed. Drop out percentage was not collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Home Care
Description: Quantitate the proportion of mothers who feel comfortable with home care of their infant at discharge
Time Frame: as for outcome 8
Population: Study closed prematurely due to poor accrual and no analysis was completed. Proportion of mothers data was not collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Readiness of Mothers to Assess Infant
Description: Monitor the readiness of mothers to assess infant on 3 to 4 hours intervals while at home
Time Frame: as for outcome 8
Population: Study closed prematurely due to poor accrual and no analysis was completed. Readiness of mothers was not assessed/collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Compliance With Pediatrician Visits
Description: Determine the compliance rate with the Johns Hopkins All Children's Hospital (JHACH) pediatrician visits.
Time Frame: as for outcome 8
Population: Study closed prematurely due to poor accrual and no analysis was completed. Compliance rate was not assessed/collected.
Arm/Group | Methadone Treatment Group | Comparison Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected throughout study participation until 12 months of age in the methadone arm. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for the Comparison Group.
Description: AEs as defined in the clinicaltrials.gov site and must meet at least one of the following:
  Possibly related to study drug, unexpected in nature or severity OR One of the following:
  Respiratory depressions, bronchospasm, angioneurotic edema, anaphylactic shock, need for respiratory support, cardiovascular compromise
  All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for the Comparison Group.
Arm/Group | Methadone Treatment Group | Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT03134703/Prot_SAP_000.pdf
  • Informed Consent Form (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT03134703/ICF_001.pdf